CLINICAL TRIAL: NCT01074697
Title: A Multinational, Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Tolerability of Palonosetron and Dexamethasone Plus Fosaprepitant or Placebo in Patients Receiving Radiotherapy and Weekly Cisplatin.
Brief Title: Efficacy of Two Antiemetic Regimens in Patients Receiving Radiotherapy and Concomitant Weekly Cisplatin
Acronym: GAND-emesis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Helsinn Healthcare SA (Industry)
Responsible Party: Principal Investigator, Christina Ruhlmann, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GAND-emesis; 2009-014691-21 (EudraCT Number)
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Nausea; Vomiting; Genital Neoplasms, Female
Keywords: Randomized Controlled Trial; Serotonin Agonists; Dexamethasone; Receptors, Neurokinin-1; Radiotherapy; Cisplatin; Prevention & control
MeSH Terms: conditions — Nausea; Vomiting; Genital Neoplasms, Female | interventions — fosaprepitant; Palonosetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fosaprepitant dimeglumine (Active Comparator)
  Interventions: Drug: Fosaprepitant dimeglumine
- Saline water (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fosaprepitant dimeglumine — Addition of fosaprepitant dimeglumine 150 mg IV single dose weekly (before chemotherapy) to dexamethasone and palonosetron.
  Other Names: Palonosetron; Dexamethasone
  Arms: Fosaprepitant dimeglumine
Drug: Placebo — Saline water
  Arms: Saline water

SUMMARY:
GAND-emesis is a multinational, randomized, double-blind, placebo-controlled, parallel-group study to investigate the efficacy and tolerability of a neurokinin1 receptor antagonist (fosaprepitant dimeglumine) in combination with an antiemetic (anti-nausea-and-vomiting) control regimen (palonosetron and dexamethasone) in patients with a gynaecological cancer diagnosis, who are scheduled to receive radiotherapy and weekly chemotherapy.

The study aims at investigating if a three-drug antiemetic regimen is superior to a two-drug regimen (standard treatment) in preventing nausea and vomiting in patients receiving radiotherapy and weekly chemotherapy. A pilot study demonstrated that approximately 50% of patients will experience nausea and vomiting when offered a two-drug antiemetic regimen, and it is expected that addition of a third drug (a neurokinin1 receptor antagonist) can increase the proportion of patients with no vomiting in the course of combined chemo-radiotherapy.

ELIGIBILITY:
Inclusion Criteria: (abbreviated)

1. The patient has a diagnosis cervical cancer.
2. The patient understands the nature and purpose of this study and the study procedures and has signed informed consent.
3. The patient is aged > 18 years.
4. The patient must be both chemo- and radiotherapy (RT) naïve. NB: previously low voltage RT or electron RT for non-melanoma skin cancers is allowed.
5. The patient is scheduled to receive fractionated radiotherapy and concomitant weekly cisplatin at a dose of ≥ 40 mg/m2 for at least five weeks.
6. Brachy therapy is scheduled to be initiated after the third cycle of weekly cisplatin, and preferentially after the fifth week of treatment.
7. Chemotherapy with an emetic risk potential of minimal or mild (up to 30%) is allowed on days 1-4 (see ref. 14).
8. The patient has a WHO Performance Status of ≤ 2.

Exclusion Criteria: (abbreviated)

1. The patient has a current malignant diagnosis other than cervical cancer, with exception of non-melanoma skin cancers.
2. The patient is aged < 18 years.
3. The patient is scheduled to receive less than five weeks of fractionated radiotherapy and concomitant weekly cisplatin.
4. Brachy therapy is planned to be initiated before the third cycle of weekly cisplatin.
5. The patient has been previously treated with radiotherapy, and/or chemotherapy, with exception of treatment with low voltage RT or electron RT for non-melanoma skin cancers .
6. The patient has a WHO Performance Status of > 2.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2010-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To compare fosaprepitant dimeglumine, palonosetron, and dexamethasone with palonosetron, dexamethasone, and placebo with respect to efficacy; the proportion of subjects with no vomiting during five weeks of radiotherapy and concomitant weekly cisplatin. | 35 days

SECONDARY OUTCOMES:
To compare the fosaprepitant dimeglumine regimen and the control regimen in terms of the proportion of subjects with complete response in the 7 days following initiation of radiotherapy and concomitant weekly cisplatin. | 7 days
To compare the fosaprepitant dimeglumine regimen and the control regimen in terms of the proportion of subjects with no significant nausea during five weeks of fractionated radiotherapy and concomitant weekly cisplatin at a dose of ≥ 40 mg/m2. | 35 days
To compare the fosaprepitant dimeglumine regimen and the control regimen with respect to complete response in the 35 days following initiation of fractionated radiotherapy and concomitant weekly cisplatin at a dose of ≥ 40 mg/m2. | 35 days
To compare the fosaprepitant dimeglumine regimen and the control regimen in terms of the proportion of subjects with no nausea during five weeks (35 days) of fractionated radiotherapy and concomitant weekly cisplatin at a dose of ≥ 40 mg/m2. | 35 days
To compare the fosaprepitant dimeglumine regimen and the control regimen in terms of the number of days to first emetic episode. | 0-35 days
To compare quality of life using the FLIE questionnaire. | 0-35 days
To compare tolerability of both regimens. | 0-35 days

CONTACTS AND LOCATIONS:
Overall Officials: Jorn Herrstedt, MD, DMSci, Study Director — Odense University Hospital; Christina Ruhlmann, MD, Principal Investigator — Odense University Hospial; Dorothy Keefe, MD, FRACP, Principal Investigator — Royal Adelaide Hospital; Petra Feyer, MD, DMSci, Principal Investigator — Vivantes Klinikum Neukölln in Berlin; Thomas Broe Christensen, MD, PhD, Principal Investigator — Herlev Hospital; Gunnar Kristensen, MD, PhD, Principal Investigator — Norwegian Radium Hospital; Henrik Roed, MD, DMSci, Principal Investigator — The Finsen Centre, Copenhagen University Hospital; Felix Hilpert, MD, DMSci, Principal Investigator — University Hospital Schleswig-Holstein; Jacob C Lindegaard, MD, Principal Investigator — Department of Oncology,Aarhus University Hospital, Aarhus, Denmark
Locations (8):
- RAH Cancer Centre, Royal Adelaide Hospital, Adelaide SA, Australia
- Denmark (4):
  - Department of Oncology, Aarhus
  - Rigshospitalet, Finsen Centret, Copenhagen
  - Herlev Hospital, Herlev
  - Department of Oncology, Odense University Hospital, Odense
- Germany (2):
  - Vivantes Klinikum Neukolln, Berlin
  - Universitatsklinikum Schleswig Holstein, Kiel
- The Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Derived] Ruhlmann CH, Christensen TB, Dohn LH, Paludan M, Ronnengart E, Halekoh U, Hilpert F, Feyer P, Kristensen G, Hansen O, Keefe D, Herrstedt J. Efficacy and safety of fosaprepitant for the prevention of nausea and emesis during 5 weeks of chemoradiotherapy for cervical cancer (the GAND-emesis study): a multinational, randomised, placebo-controlled, double-blind, phase 3 trial. Lancet Oncol. 2016 Apr;17(4):509-518. doi: 10.1016/S1470-2045(15)00615-4. Epub 2016 Mar 4. PMID 26952945